CLINICAL TRIAL: NCT06971068
Title: Endovenous Vacuum-assisted Laser Ablation (VALA) in the Treatment of Large Saphenous Veins (> 15 mm)
Brief Title: Vacuum-assisted Laser Ablation (VALA) for Treatment of Large Saphenous Veins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center Of Phlebology (Network)
Responsible Party: Principal Investigator, Dmitrii Alekseev, Director, Center Of Phlebology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CenterPhlebology
Record Dates: First submitted 2025-05-02; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Varicose Veins
Keywords: Vacuum-assisted Laser Ablation; large saphenous veins; varicose veins; EVLA
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial 2ring fiber (Active Comparator): Refluxing GSV/SSV treated with endovenous laser ablation using ELVeS Radial 2ring fiber
  Interventions: Procedure: Procedure: EVLA
- Radial 2ring Pro fiber (Active Comparator): Refluxing GSV/SSV treated with endovenous laser ablation using ELVeS Radial 2ring Pro fiber
  Interventions: Procedure: Procedure: VALA

INTERVENTIONS:
Procedure: Procedure: EVLA — Great or small saphenous vein occlusion with endovenous laser ablation using ELVeS Radial 2ring fiber
  Arms: Radial 2ring fiber
Procedure: Procedure: VALA — Great or small saphenous vein occlusion with endovenous laser ablation using ELVeS Radial 2ring Pro fiber
  Arms: Radial 2ring Pro fiber

SUMMARY:
Endovenous thermal ablation (EVTA), including radiofrequency ablation (RFA) and endovenous laser ablation (EVLA), is considered the main method for the treatment of symptomatic truncal vein reflux. However, there are controversial data concerning their efficacy and safety in ablating large saphenous veins because of high risk of heat-induced thrombosis (EHIT), incomplete ablation and recanalization.1-5 The use of vacuum evacuation of the remaining intraluminal blood during endovenous laser ablation allows to decrease the risk of intraoperative (carbonization and destruction of the fiber lens) and postoperative complications (EHIT, hyperpigmentation, "string" feeling) and leads to reduction of recovery because of short period of vein resorption. The aim of the study is to evaluate the safety and effectiveness of endovenous thermal ablation with or without vacuum evacuation for the treatment of incompetent large saphenous veins (>15 mm).

DETAILED DESCRIPTION:
Preoperatively all patients should be examined in a standing position clinically and with duplex ultrasound (DUS) marking of the diameters of the target great saphenous veins (GSV) or small saphenous veins (SSV) at the following levels:

* great saphenous vein: saphenofemoral junction (SFJ), vein ectasia below the SFJ by 3 cm, upper third of the thigh, middle third of the thigh, lower third of the thigh, upper third of the leg, middle third of the leg, lower third of the leg;
* small saphenous vein: saphenopopliteal junction (SPJ), ectasia below the SPJ by 3 cm, upper third of the leg, middle third of the leg, lower third of the leg.

It is recommended to calculate the required linear energy density (LEED) per centimeter of vein length using the following formula depending on the level of measurement of the target vein diameter: LEED=d*k, where LEED is the linear energy density (J/cm), "d" is the vein diameter (mm), "k" is the coefficient based on the measurement level: upper half of the thigh - 10, lower half of the thigh - 8, upper half of the leg - 6, lower half of the leg - 4.

Under local anesthesia, the target vein is punctured and the introducer is then installed. For the first group of patients (ELVeS Radial 2ring fiber), there is no need for preliminary preparation of the fiber. For the second group (ELVeS Radial 2ring Pro fiber), it is recommended to fill the ELVes Radial 2ring Pro catheter with a pre-prepared heparin solution (200 ml 0.9% Na Cl + 1 ml (5000) heparin) before use. Passing the fiber and installing it in the orifice of the target vein. Performing tumescent anesthesia (1000 ml 0.9% NaCl, 10 ml 2% lidocaine, 0.25 ml 0.1% adrenaline, 56 ml 4% sodium bicarbonate at room temperature) with recording the volume of the solution used. Performing EVLA with recording the parameters at different levels (power, extraction rate). When performing laser obliteration in patients of the second group, the ELVeS Radial 2ring Pro fiber catheter is connected to a vacuum suction using a high-pressure line to evacuate residual blood from the lumen of the vein during EVLA. Compression underwear of class 2 according to RAL or class 3 according to ASQUAL (23-32 mm Hg).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Varicose veins of the lower extremities with clinical class C2-C6 with a diameter of the GSV or SSV ≥ 15 mm in a standing position
* Informed consent

Exclusion Criteria:

* pregnancy or lactation
* malignant neoplasms
* inability or unwillingness of any patient to wear compression stockings
* hypersensitivity to lidocaine
* concomitant diseases: diabetes mellitus, bronchial asthma, severe liver and kidney diseases, acute thrombosis and thrombophlebitis, skin and/or soft tissue infection, infectious diseases, obliterating peripheral arteriosclerosis, diabetic angiopathy, heart defects requiring surgical intervention, fever, toxic hyperthyroidism, obesity, tuberculosis, sepsis, blood cell composition disorder, all diseases requiring bed rest, heart disease with decompensation, known hereditary thrombophilia
* period after treatment for alcohol addiction
* sedentary lifestyle
* history of acute deep vein thrombosis
* history of superficial thrombophlebitis
* history of drug or other addiction
* use of oral contraceptives or other hormonal drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Occlusion of the treated GSV/SSV | One day, 2 weeks, one month, 3 months and 6 months post treatment
  Obliteration of varicose vein along the treated segment of the GSV/SSV measured using ultrasound (US) examination

SECONDARY OUTCOMES:
Pain score and use of painkillers | One day, 2 weeks, one month, 3 months and 6 months post treatment
  A questionnaire including the Numeric Rating Scale (NRS) of pain is filled in by the patient. It is a numeric scale from 0 (no pain) to 10 (worst imaginable pain).
Clinical status | 2 weeks, one month, 3 months and 6 months post treatment
  CEAP classification. The CEAP classification is a common descriptive platform for the reporting of diagnostic information in chronic venous disease, as well as a tool for regular patient documentation and management. The clinical component indicates disease severity, ranging from none (0 points) to active ulcers (6 points). The etiologic component denotes the venous disease as congenital, primary, or secondary in nature. The anatomic classification pinpoints the veins involved as superficial, deep, or perforating. The pathophysiologic classification identifies the presence of reflux in the superficial,communicating, or deep systems, as well as the existence of outflow obstruction.
Severity of chronic venous diseases | 2 weeks, one month, 3 months and 6 months post treatment
  Venous Clinical Severity Score (VCSS). The VCSS includes 9 hallmarks of venous disease, each scored on a severity scale from 0 to 3.
Health related quality of life | one month, 3 months and 6 months post treatment
  A questionnaire Chronic Venous Insufficiency Questionnaire (CIVIQ 20) is filled in by the patient. The CIVIQ comprises 20 questions in four quality-of-life domains: physical, psychological, social, and pain.The result ranges from 0 to 100.
Histological picture of the treated vein | 2 weeks, one month, 3 months post treatment
  A time period of connective tissue transformation of the vein wall and its lysis assessed by histochemical analysis (Picro-Mallory, Martius-Scarlet-Blue, Fuchsin-Miller)
Number of patients with adverse events | One day, 2 weeks, one month, 3 months and 6 months post treatment
  Major complications: superficial and deep venous thrombosis including EHIT, nerve injury, skin burns, and subcutaneous infections. Minor complications: ecchymosis and hyperpigmentation
Severity of hyperpigmentation | 2 weeks, one month, 3 months and 6 months post treatment
  Skin tone estimated using the Pantone SkinTone Guide and compared with an unchanged area of skin

CONTACTS AND LOCATIONS:
Locations (8):
- Belarus (3):
  - Clinic in Uruchye, Minsk
  - Merci clinic, Minsk
  - SANTE clinic, Minsk
- Center Of Phlebology, Bishkek, Chuy Region, Kyrgyzstan
- Russia (3):
  - Laser Surgery Center, Moscow
  - Innovative vascular centre, Saint Petersburg
  - Derzhavin Tambov State University, Tambov
- Clinic of Modern Phlebology "VarikozOFF", Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Yes
The study data are available to all investigators in the chronic vein disease registry
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 15 March 2025 to 15 February 2026

REFERENCES:
- [Background] Van der Velden SK, Lawaetz M, De Maeseneer MG, Hollestein L, Nijsten T, van den Bos RR; Members of the Predictors of Endovenous Thermal Ablation Group. Predictors of Recanalization of the Great Saphenous Vein in Randomized Controlled Trials 1 Year After Endovenous Thermal Ablation. Eur J Vasc Endovasc Surg. 2016 Aug;52(2):234-41. doi: 10.1016/j.ejvs.2016.01.021. Epub 2016 Mar 16. PMID 26994834
- [Background] Sufian S, Arnez A, Labropoulos N, Lakhanpal S. Endovenous heat-induced thrombosis after ablation with 1470 nm laser: Incidence, progression, and risk factors. Phlebology. 2015 Jun;30(5):325-30. doi: 10.1177/0268355514526588. Epub 2014 Mar 7. PMID 24609619
- [Background] Bontinis V, Bontinis A, Koutsoumpelis A, Potouridis A, Giannopoulos A, Rafailidis V, Chorti A, Ktenidis K. Endovenous thermal ablation in the treatment of large great saphenous veins of diameters > 12 mm: A systematic review meta-analysis and meta-regression. Vasc Med. 2023 Oct;28(5):449-457. doi: 10.1177/1358863X231183997. Epub 2023 Jul 17. PMID 37458188
- [Background] Elboushi A, Elsherbeni M, Gameel AM, et al. The 1470 radial endovenous laser ablation of the great saphenous vein larger than 12 mm: Is it a good option? A single-center expe-rience? Egyptian J Surg 2019; 38: 136-141.
- [Background] Dabbs EB, Mainsiouw LE, Holdstock JM, Price BA, Whiteley MS. A description of the 'smile sign' and multi-pass technique for endovenous laser ablation of large diameter great saphenous veins. Phlebology. 2018 Sep;33(8):534-539. doi: 10.1177/0268355517734480. Epub 2017 Sep 28. PMID 28956693